CLINICAL TRIAL: NCT00176332
Title: Impact of Three Months of Rosuvastatin Treatment on Peripheral Endothelial Function, Inflammatory Markers in the Blood and the Skeletal Muscle and on Postnatal Vasculogenesis in Patients With Severe Chronic Heart Failure
Brief Title: Impact of Rosuvastatin on Endothelial Function and Inflammation in Patients With Chronic Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: AstraZeneca (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 121/2003
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2007-08-01 (Estimated); Status verified 2007-07

CONDITIONS: Heart Failure
Keywords: chronic heart failure; rosuvastatin; endothelial function; skeletal muscle
MeSH Terms: conditions — Heart Failure | interventions — Rosuvastatin Calcium

INTERVENTIONS:
Drug: rosuvastatin

SUMMARY:
Statin therapy has been shown to efficiently reduce mortality in patients with coronary artery disease and myocardial infarction, partially as a result of the lipid-lowering properties of statins. However, especially the pleiotropic effects of statins, e.g. their anti-inflammatory and anti-oxidative properties, might be of interest in the treatment of patients with chronic heart failure that are limited in their exercise capacity due to alterations of the skeletal muscle and peripheral endothelial dysfunction.

Aim of this trial is therefore to assess the effects of three months of rosuvastatin treatment on markers of inflammation and oxidative stress in the skeletal muscle and the blood, on postnatal vasculogenesis, and endothelial function of the radial artery in patients with severe chronic heart failure.

DETAILED DESCRIPTION:
A total of 40 patients with severe chronic heart failure are prospectively randomized to either 3 months of rosuvastatin or placebo treatment.

Before and after the intervention period maximal exercise capacity is measured by ergospirometry and endothelial function is determined by high-resolution A-mode ultrasound. Skeletal muscle biopsies are obtained at begin and after 3 months and are analyzed for inflammatory markers, measures of oxidative stress and vasculogenesis. Blood samples are assessed with regard to markers of inflammation and oxidative stress as well.

ELIGIBILITY:
Inclusion Criteria:

* chronic heart failure (NYHA class III or IV)
* peak oxygen uptake <20 mL/min/kg body weight
* left ventricular ejection fraction <30 %
* left ventricular end-diastolic diameter >55 mm
* stable medication within the last 4 weeks

Exclusion Criteria:

* elevated GOT and GPT levels as a sign of hepatic dysfunction
* elevated creatinine levels as a sign of renal dysfunction
* insulin-dependent diabetes mellitus
* arterial hypertension
* muscle disease or elevated CK levels
* treatment with fibrates
* co-treatment with drugs that are metabolized by Cyp3A4
* diseases that disallow a participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-03; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Inflammation in the blood and the skeletal muscle
Vasculogenesis
Endothelial function of the radial artery

SECONDARY OUTCOMES:
Peak oxygen uptake
Left ventricular function

CONTACTS AND LOCATIONS:
Overall Officials: Rainer P Hambrecht, MD, Principal Investigator — University of Leipzig, Heart Center, Department of Internal Medicine / Cardiology
Locations (1):
- University of Leipzig, Heart Center, Department of Internal Medicine / Cardiology, Leipzig, Saxony, Germany